CLINICAL TRIAL: NCT01630083
Title: A Randomized Phase II Multicenter, Open-Label Study Evaluating the Efficacy and Safety of IMAB362 in Combination With the EOX (Epirubicin, Oxaliplatin, Capecitabine) Regimen as First-Line Treatment of Patients With CLDN18.2-Positive Advanced Adenocarcinomas of the Stomach, the Esophagus or the Gastroesophageal Junction
Brief Title: Efficacy and Safety of IMAB362 in Combination With the EOX Regimen for CLDN18.2-positive Gastric Cancer
Acronym: FAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: GM-IMAB-001-03; 2011-005285-38 (EudraCT Number); 8951-CL-0202 (Other: Astellas)
Record Dates: First submitted 2012-06-19; First posted 2012-06-28 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: CLDN18.2-positive Adenocarcinoma of the Gastroesophageal Junction; CLDN18.2-positive Adenocarcinoma of Esophagus; CLDN18.2-positive Gastric Adenocarcinoma
Keywords: IMAB362; ASP8951; zolbetuximab
MeSH Terms: interventions — Epirubicin; Oxaliplatin; Capecitabine; zolbetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EOX Treatment (Active Comparator): Participants will receive up to 8 cycles of epirubicin, oxaliplatin and capecitabine (EOX) chemotherapy treatment alone (50 mg/m^2 epirubicin intravenously on day 1 of each cycle, 130 mg/m^2 oxaliplatin intravenously on day 1 of each cycle, 625 mg/m^2 capecitabine orally twice daily on days 1 to 21 of each cycle). The first dose of capecitabine to be taken in the evening of day 1.
  Interventions: Drug: epirubicin; Drug: oxaliplatin; Drug: capecitabine
- EOX+zolbetuximab 800/600 mg/m^2 (Experimental): Participants will received up to 8 cycles of EOX chemotherapy treatment in combination with zolbetuximab administered as loading dose of 800 mg/m^2 intravenously on day 1 of cycle 1 followed by 600 mg/m^2 intravenously on day 1 of each subsequent cycle. Zolbetuximab to be administered prior to EOX chemotherapy. After completion of the EOX treatment phase, participants will be permitted to continue zolbetuximab monotherapy (600 mg/m^2 every 3 weeks to be administered intravenously as a 2-hour infusion) until progressive disease (PD), withdrawal of consent or unacceptable toxicity. PD per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study, an absolute increase of at least 5mm must also be demonstrated, unequivocal progression of existing non-target lesions and appearance of one or more new lesions is considered progression.
  Interventions: Drug: epirubicin; Drug: oxaliplatin; Drug: capecitabine; Drug: zolbetuximab
- EOX+zolbetuximab 1000 mg/m^2 (Experimental): Participants will receive up to 8 cycles of EOX chemotherapy treatment in combination with zolbetuximab 1000 mg/m^2 intravenously on day 1 of each cycle. Zolbetuximab to be administered prior to EOX chemotherapy. After completion of the EOX treatment phase, participants will be permitted to continue zolbetuximab monotherapy (1000 mg/m^2 every 3 weeks administered intravenously as a 2-hour infusion ) until PD, withdrawal of consent or unacceptable toxicity.
  Interventions: Drug: epirubicin; Drug: oxaliplatin; Drug: capecitabine; Drug: zolbetuximab

INTERVENTIONS:
Drug: epirubicin — Epirubicin will be administered at a dose of 50 mg/m^2 as a 15-minute intravenous infusion on day 1 of each cycle.
Drug: oxaliplatin — Oxaliplatin will be administered at a dose of 130 mg/m^2 as a 2-hour intravenous infusion on day 1 of each cycle.
Drug: capecitabine — The daily dose of capecitabine will be 1250 mg/m^2. Capecitabine tablets to be given once daily at a dose of 625 mg/m^2 orally in the evening of day 1 of each cycle and twice daily at a dose of 625 mg/m^2 orally on days 2 to 21 of each cycle; the morning dose of capecitabine on day 1 of each cycle to be omitted due to administration of zolbetuximab, epirubicin and oxaliplatin.
Drug: zolbetuximab — Two different formats of zolbetuximab, comprising different strengths, to be provided. Vials contained 22 mg or 105 mg of zolbetuximab. Prior to administration, zolbetuximab will be reconstituted with 1.1 mL (22 mg zolbetuximab vials) or 5.0 mL (105 mg zolbetuximab vials) water for injection, which will result in a concentration of 20 mg/mL zolbetuximab. The extractable volume per vial will be 1 mL (for 22 mg zolbetuximab vials) or 5 mL (for 105 mg zolbetuximab vials). The reconstituted solution will be further diluted with sodium chloride 0.9% to a final concentration of 2 mg/mL zolbetuximab. Zolbetuximab will be administered as an intravenous infusion over 2 to 3 hours.
  Other Names: IMAB362
  Arms: EOX+zolbetuximab 1000 mg/m^2; EOX+zolbetuximab 800/600 mg/m^2

SUMMARY:
The purpose of the trial is to assess the therapeutic effects and the safety profile of IMAB362 combined with EOX (epirubicin, oxaliplatin, capecitabine) as first-line treatment for patients with advanced adenocarcinoma of the stomach, the esophagus or the gastroesophageal junction compared to EOX alone.

Furthermore, sufficient binding of IMAB362 to the target cells is necessary for antitumoral activity. Thus, two dose levels ensuring a serum level above the in vitro predicted clinical efficacy threshold will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach, the esophagus or the gastroesophageal junction
* Inoperable locally advanced disease or resections with R2 outcome or recurrent or metastatic disease.
* CLDN18.2 expression confirmed by immunohistochemistry in paraffin embedded tumor tissue sample.
* Measurable and/or non-measurable disease as defined according to RECISTv1.1
* Age ≥ 18 years
* Written Informed Consent Form
* ECOG performance status (PS) 0-1
* Life expectancy > 3 months
* HER2/neu negative patients and patients with HER2/neu positive status but not eligible to trastuzumab therapy in discretion of the investigator.
* Adequate cardiac, hepatic, renal, hematologic function.

Exclusion Criteria:

* Prior severe allergic reaction or intolerance to a monoclonal antibody, to the chemotherapeutics used in this study or any excipient in the respective formulations.
* Previous chemotherapy for advanced disease.
* Previous perioperative chemotherapy with curative intention within 6 months of start of study treatment. If interval is longer than 6 months (counted from the stop date of the perioperative chemotherapy), patients are allowed.
* Known HIV infection or known symptomatic hepatitis (A, B, C).
* Symptomatic cerebral metastases.
* Pregnancy or breastfeeding.
* Previous treatments with maximum cumulative doses of epirubicin > 500 mg/m² and/or other anthracyclines and anthracenediones.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2012-07-19 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to the data cut-off date of 31JAN2019; maximum time on follow-up was, 68.2, 47.2 & 59.6 months in the EOX, EOX+Zolbetuximab 600 mg, and EOX+Zolbetuximab 1000 mg treatment groups respectively.
  PFS is defined as the time from randomization to the first observation of disease progression (based on central reading) or death from any cause (as assessed by the independent reviewer). Participants without documented progression or death will be censored as of the last tumor evaluation determining lack of progression.
Number of Participants with Adverse Events (AEs) | From the first dose of study drug administration up to 30 days after the last study medication administration (up to 1791 days).
  An AE is defined as any unintended or undesirable, noxious or pathological change, compared to pre-existing conditions, experienced by a participant during a clinical study or the follow-up period, regardless of relationship to study medication. Treatment-emergent adverse event (TEAE) are those AEs that started or worsened after the first dose of study medication.

SECONDARY OUTCOMES:
Clinical PFS | From randomization to the data cut-off date of 31JAN2019; maximum time on follow-up was, 68.2, 47.2 & 59.6 months in the EOX, EOX+Zolbetuximab 600 mg, and EOX+Zolbetuximab 1000 mg treatment groups respectively.
  Clinical PFS (CPFS) is defined as the time from randomization to the first observation of disease progression, either confirmed by computed tomography (CT) scans or by clinical evaluation, or death from any cause (as assessed by the independent reviewer with clinical PD considered as an event). Participants without documented progression or death will be censored as of the last tumor evaluation determining lack of progression.
Overall Survival Rate at 12 Months | Up to 12 months
  Overall survival rate at 12 months after therapy initiation is defined as a proportion of participants alive after 12 months from first dose of any study drug.
Overall Survival (OS) | From randomization to the data cut-off date of 31JAN2019; maximum time on follow-up was, 68.2, 47.2 & 59.6 months in the EOX, EOX+Zolbetuximab 600 mg, and EOX+Zolbetuximab 1000 mg treatment groups respectively.
  OS is defined as the time from randomization to death from any cause or last contact (if alive).
Time to Progression (TTP) | From randomization to the data cut-off date of 31JAN2019; maximum time on follow-up was, 68.2, 47.2 & 59.6 months in the EOX, EOX+Zolbetuximab 600 mg, and EOX+Zolbetuximab 1000 mg treatment groups respectively.
  TTP is defined as the time from randomization to the first observation of disease progression (based on central reading as assessed by the investigator reviewer). Participants without documented progression will be censored as of the last tumor evaluation determining lack of progression.
Objective Tumor Response Rate (ORR) | Up to week 94
  ORR is defined as the fraction of participants with a complete response (CR) or partial response (PR), according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (as assessed by the investigator reviewer). CR according to RECIST v1.1 is defined as the disappearance of all target lesions, any pathological lymph node must have reduction in short axis to < 10 mm, disappearance of all non-target lesions and normalization of tumor marker level should occur as well as no simultaneous appearance of new lesions. PR according to RECIST v1.1 is defined as at least 30% decrease in the sum of the longest diameter of target lesions, taking as reference the screening sum longest diameter and no simultaneous increase in the size of any lesion or the appearance of new lesions.
Disease Control Rate (DCR) | Up to week 94
  DCR is defined as the fraction of participants with CR or PR or stable disease (SD) according to RECIST v1.1 (as assessed by the investigator reviewer). SD according to RECIST v1.1 is defined as neither sufficient shrinkage to qualify for PR or CR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter recorded since treatment started, measurements must meet the SD criteria at least once after study entry at a minimum interval not less than 6 weeks, no simultaneous increase in the size of any lesion or the appearance of new lesions should occur, evaluable lesions must remain stable or regress for this category.
Duration of Response (DOR) | From randomization to the data cut-off date of 31JAN2019; maximum time on follow-up was, 68.2, 47.2 & 59.6 months in the EOX, EOX+Zolbetuximab 600 mg, and EOX+Zolbetuximab 1000 mg treatment groups respectively.
  DOR will be determined as the time when criteria for CR or PR are first met until the first date that recurrent or progressive disease or death occurs (as assessed by the independent reviewer).

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (48):
- Bulgaria (5):
  - Site BUL004, Plovdiv
  - Site BUL001, Sofia
  - Site BUL003, Sofia
  - Site BUL005, Sofia
  - Site BUL002, Varna
- Czechia (2):
  - Site CZE002, Olomouc
  - Site CZE001, Znojmo
- Germany (10):
  - Site GER012, Bielefeld
  - Site GER029-01, Bochum
  - Site GER029, Bochum
  - Site GER010, Dresden
  - Site GER001, Essen
  - Site GER017, Frankfurt
  - Site GER005, Halle
  - Site GER020, Leipzig
  - Site GER016, Münster
  - Site GER013, Pinneberg
- Latvia (2):
  - Site LAT001, Liepāja
  - Site LAT002, Riga
- Russia (17):
  - Site RUS011, Arkhangelsk
  - Site RUS016, Bryansk
  - Site RUS006, Chelyabinsk
  - Site RUS007, Ivanovo
  - Site RUS009, Kursk
  - Site RUS001, Moscow
  - Site RUS002, Obninsk
  - Site RUS023, Omsk
  - Site RUS014, Orenburg
  - Site RUS012, Oryol
  - Site RUS005, Pyatigorsk
  - Site RUS019, Ryazan
  - Site RUS003, Saint Petersburg
  - Site RUS010, Saint Petersburg
  - Site RUS015, Saint Petersburg
  - Site RUS017, Veliky Novgorod
  - Site RUS013, Yaroslavl
- Ukraine (12):
  - Site UKR003, Dnipropetrovsk
  - Site UKR001, Donetsk
  - Site UKR002, Donetsk
  - Site UKR008, Ivano-Frankivsk
  - Site UKR005, Kharkiv
  - Site UKR007, Kyiv
  - Site UKR006, Lviv
  - Site UKR015, Poltava
  - Site UKR004, Simferopol
  - Site UKR011, Sumy
  - Site UKR010, Uzhhorod
  - Site UKR009, Zaporizhia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/GM-IMAB-001-03/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=25768&tenant=MT_AST_9011